CLINICAL TRIAL: NCT04679142
Title: Baclocur® Post-Authorisation Safety Study in Real-life Settings in France
Acronym: BACLOLIFE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ethypharm (Industry)
Responsible Party: Sponsor
Other Study IDs: ALP2011007/005; ID-RCB: 2020-A00722-37 (Other: ANSM FRANCE)
Record Dates: First submitted 2020-12-07; First posted 2020-12-22 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Baclofen

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients starting a treatment with Baclocur®: Baclofen(Baclocur®) 10mg, 20mg, 30mg, 40mg.
  Interventions: Drug: Baclofen Tablets

INTERVENTIONS:
Drug: Baclofen Tablets — Enrolled patients will receive treatment and evaluations for their disease as determined by their physicians in accordance with local standard of care. Visits will be scheduled by their physician according to patient-specific needs and national clinical practice.
  Other Names: Baclocur®

SUMMARY:
The overall goal of the study is to further characterize the risks and the safety profile of Baclocur® in real life settings, over a 12-month follow-up period.

DETAILED DESCRIPTION:
This is a prospective, multicenter, non-comparative non-interventional post-authorisation safety study (PASS) conducted in France. There will be no experimental intervention utilized. Enrolled patients will receive treatment and evaluations for their disease as determined by their physicians in accordance with local standard of care. Visits will be scheduled by their physician according to patient-specific needs and national clinical practice.

For purposes of this study, physicians will be requested to record information on enrolled patients at the time of study enrolment (baseline), and then to conduct follow-up patient visits based on their usual practice for a period of 12 months following Baclocur® initiation.

At study end, further investigations on patients confirmed as lost to follow-up (LFU) will be performed through the use of the French medico-administrative database called the Système National des Données de Santé (SNDS). The goal will be to determine their vital status and collect relevant treatment and safety data over the studied period to further assess the safety of Baclocur®. A probabilistic approach using relevant matching variables (e.g. gender, year of birth, date of Baclocur prescription, department of care) will be used to retrieve these SNDS data of interest.

The patient study enrolment period is expected to be approximately of 3 years. Accounting for the 12 months follow-up period per patient, the full study field duration is expected to be approximately of 4 years. One additional year will be needed before the SNDS matching is performed, taken into account the delay required for the SNDS to be updated. With the final analysis and final clinical study report, this will lead to a total study duration of approximately 6 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 or more;
2. Initiating a treatment with Baclocur®;
3. Informed and having agreed to participate in the study;
4. Covered by healthcare insurance.

Exclusion Criteria:

1. Current participation in a clinical trial;
2. Previous treatment with baclofen/Baclocur®;
3. Patient deprived of liberty by a judicial or administrative decision, or who is under a measure of legal protection (e.g. guardianship or curatorship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients starting a treatment with Baclocur®. Patients having already taken Baclocur®/baclofen in the past are not eligible; only treatment-naïve patients are eligible.
Sampling Method: Probability Sample
Enrollment: 975 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious adverse events (SAE) | 12-month follow-up period
  To estimate the incidence of serious adverse events (SAE)

SECONDARY OUTCOMES:
Incidence of all adverse events over the 12-month follow-up | 12-month follow-up period
  Incidence of all adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Henri-Jean Aubin, MD, Ph.D, Principal Investigator — Hospital Paul Brousse Villejuif France
Locations (1):
- CHU Dijon, Dijon, France